CLINICAL TRIAL: NCT04192539
Title: The Prospect of Using Serum Taurine Level as a Potential Biomarker for Early Detection of Colorectal Carcinoma and Its Correlation With Other Prognostic Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: FWA00007284
Record Dates: First submitted 2019-12-07; First posted 2019-12-10 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Taurine in Cancer Colon

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator)
  Interventions: Diagnostic Test: Taurine
- Inflammation (Active Comparator)
  Interventions: Diagnostic Test: Taurine
- Benign group (Active Comparator)
  Interventions: Diagnostic Test: Taurine
- Malignant group (Active Comparator)
  Interventions: Diagnostic Test: Taurine

INTERVENTIONS:
Diagnostic Test: Taurine — Serum taurine was determined by High Performance Liquid Chromatography (HPLC) according to the pre-column extraction and derivatization methodology of McMahon et al. In the present work, we use Shimadzu HPLC model LC-10AT

SUMMARY:
Serum taurine results in this study showed that, besides CRC biomarkers; it is most attractive, more precious and more accurate early biomarker for early detecting of any malignant change which may led to CRC by other mean it is the most sensitive and more specific tumor marker for CRC. As a result, we can recommend measuring its level regularly with other prognostic tumor biomarkers and screening examination for all people with abdominal and gastrointestinal problems and for precancerous patients as a pre-early biomarker for colorectal carcinoma. So, it needs further studies to confirm that observations on large scale of population as it obvious the small sample size in early stage and lack data due to limited financial resources and it needs more efforts to collect first and precancerous stages patients.

DETAILED DESCRIPTION:
Two-hundred and fifty Egyptian patients (males and females) who attended National Cancer Institute, Cairo university; most of them were referred from private clinics and non-specialized hospitals, complain with abdominal troubles and gastrointestinal problems and bleeding per rectum, after full investigation, clinical examination, biochemical analysis, screening examination according to their cases (Ultra sound, CT or endoscopy either rectal or colonoscopy) and histopathological examination, we choose 'after their approval' one-hundred patients and six which diagnosed as CRC patients aged (19-69 years old) and excluded the others from participated in these studies because they diagnosed as non-colonic diseases like; Irritable colon, Gastroenteritis, Pancreatitis, Liver flexure or Chronic cholecystitis. According to Histopathological architecture, we divided patients to:

1. Inflammatory group number=7.
2. Benign tumor group number=8 which was assessed preoperatively and postoperatively.
3. Malignant tumor group number=91 Lastly, ten health volunteers were enrolled as a frank control. For all included subjects, the measured biochemical analysis were CBC, ALT, AST, Albumin, Total Bilirubin, Creatinine, Blood urea, Sodium, Potassium, CEA, CA19.9 and Taurine.

ELIGIBILITY:
Inclusion Criteria:

Patients complain of abdominal troubles and gastrointestinal problems and bleeding per rectum

Exclusion Criteria:

Patients refusal,non-colonic diseases like; Irritable colon, Gastroenteritis, Pancreatitis, Chronic cholecystitis

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
serum taurine levels | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: No